CLINICAL TRIAL: NCT02866201
Title: Etiological Diagnosis of Traveler's Diarrhoea
Acronym: DIAVOY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-48
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Traveler's Diarrhoea
Keywords: Turista

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient suffering from traveler's diarrhoea (Experimental): Patient suffering form traveler's diarrhoea during a stay (up to 3 months) outside metropolitan France
  Interventions: Other: Rectal swab

INTERVENTIONS:
Other: Rectal swab

SUMMARY:
Traveler's diarrhoea or turista is the most common disease in travelers. It has been reported based on studies in 20 to 60% of travelers, depending among other conditions and travel destinations. Currently, less than 30% of the etiology of diarrhoea is identified by bacteriological v,irological and parasitology traditional techniques. This ignorance of the diarrhoea etiology causes difficulties in the establishment of a specific and rapid management in this extremely common condition and having a significant cost to society. Technological advances in laboratory diagnosis, such as quantitative real-time Polymerase Chain Reaction (PCR), can allow us now to improve the etiological diagnosis of traveler's diarrhoea using simple rectal swabs.

So, the principal objective of this study is to assess the efficacy of a new diagnosis strategy in order to establissh the etiological diagnosis of traveler's diarrhoea. The hypothesis consists in improving the number of patients with a confirmed etiological diagnosis of traveler's diarrhoea by 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patient leaving for a trip outside France for a period (not exceeding 3 months)
* Patient who get seen by Travel information Service at hospital before departure.
* Adult patients (> 18 years).
* Patient who freely signed the written informed consent
* Patient affiliated to a social security regime. Exclusion criteria
* Minor patient (<18 years)
* Pregnant or nursing woman.
* Adult patient under guardianship.
* Patient deprivated with liberty under court order.
* Patient refusing to sign the wrtten consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2013-09-15 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a confirmed etiological diagnosis of traveler's diarrhoea | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided